CLINICAL TRIAL: NCT02664675
Title: Comparison of Cytokines Production and Cellular Recruitment in Gingival Crevicular Fluid (GCF) and Granulation Tissue From Periodontitis, Peri-implantitis and Healthy Patients Leading to Activation of Osteoclasts and Bone Resorption
Brief Title: Cellular and Molecular Inflammatory Mechanisms Leading to Bone Resorption in Peri-implantitis Vs Periodontitis
Acronym: DUOROPA
Status: Completed | Type: Observational
Sponsor: University of Paris 5 - Rene Descartes (Other)
Collaborators: Dentsply Sirona Implants and Consumables (Industry)
Responsible Party: Principal Investigator, Marjolaine Gosset, Associate professor in Periodontology, Faculty of dental surgery, University of Paris 5 - Rene Descartes
Other Study IDs: D-2013-003
Record Dates: First submitted 2014-04-25; First posted 2016-01-27 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Peri-Implantitis; Periodontitis
MeSH Terms: conditions — Peri-Implantitis; Periodontitis | interventions — Crown Lengthening

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — Gingiva samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Periimplantitis: patients formerly treated with a non surgical procedure without antibiotics with at least one functional dental implant with at least on pocket deeper than 5 mm with bleeding on probing and radiographical alveolar bone loss.
  These patient will be treated by open flap debridement nd the granulation tissue xill be harvested for analysis.
  Interventions: Procedure: Open Flap Debridement
- Periodontitis: patients formerly treated with a non surgical procedure without antibiotics for a generalized severe chronic periodontitis (in accord to Armitage 2009) and needing a resective surgical procedure (periodontal pockets deeper than 5 mm with bleeding on probing) These patient will be treated by open flap debridement nd the granulation tissue xill be harvested for analysis.
  Interventions: Procedure: Open Flap Debridement
- Healthy patient: healthy patients needing crown lengthening allowing collection of gingival explants
  Interventions: Procedure: Crown lengthening

INTERVENTIONS:
Procedure: Crown lengthening — After a local anesthesia, gingival tissue is removed around the teeth to extend the length of the crown for aesthetic or prosthetic matter.
  Groups: Healthy patient
Procedure: Open Flap Debridement — After local anesthesia, intra-sulcular incisions are done and a flap is released to access to the intra-bony defect.
  Granulation tissue is removed and carefully laid aside for further analysis. Interrupted sutures are done to close the flap.
  Groups: Periimplantitis; Periodontitis

SUMMARY:
Recent data found that peri-implantitis may differ from periodontitis at the histological level in terms of extent and composition of the cellular components. From human biopsies, it has been shown a deeper apical extension of the inflammatory cell infiltrate and a larger proportion of granulocytes and macrophages in peri-implantitis lesions compared to periodontitis lesions. Following experimental peri-implantitis, it has been observed a continuing bone loss around dental implants after ligature removal; whereas, such a progression was not observed around teeth after cessation of the experimental periodontitis. The factors influencing the recruitment and the activation of osteoclasts in both diseases have not been compared yet.

Hypothesis : The more rapid and more severe alveolar bone destruction occurring in peri-implantitis compared to periodontitis is due at least in part to differences in the inflammatory process in these diseases.

Aim: to study the cytokine profile produced by gingival explants from periodontitis or peri-implantitis sites and to test the consequences on alteration of bone remodelling activity using in vitro approach.

Materials and methods The investigators will establish a collection of human gingival samples from patients undergoing surgical treatment of periodontitis or peri-implantitis. The investigators will test pro-inflammatory cytokines and chemokines release and consequences on osteoclast differentiation and activity.

ELIGIBILITY:
Inclusion Criteria:

* Beneficiary by national health insurance
* Age: over 18 year-old
* Non smoking
* Good health

  ---For the periimplantitis group:
* patients formerly treated with a non surgical procedure without antibiotics with at least one functional dental implant with at least on pocket deeper than 5 mm with bleeding on probing and radiographical alveolar bone loss.

  ---For the periodontitis group:
* patients formerly treated with a non surgical procedure without antibiotics for a generalized severe chronic periodontitis (in accord to Armitage 2009) and needing a resective surgical procedure (periodontal pockets deeper than 5 mm with bleeding on probing)

  ---For the healthy group:
* patients with good health without periodontal or peri implant disease needing gingivectomy (crown lengthening, esthetic surgery)

Exclusion Criteria:

* Smokers
* Patients treated with antibiotics or NSAID during the last 3 months
* Patients suffering from a chronic infectious, inflammatory or auto-immune disease (non equilibrated diabetes mellitus, rheumatoid arthritis, spondylarthrosis, Gougerot-Sjögren, Crohn, Behcet, Horton, obesity, chronic end renal disease, cardiopathies....)
* Pregnant women
* For the healthy group : bleeding on probing on the site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated in periodontology department of Hospital Rotschild or Charles Foix
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2014-04; Primary Completion 2015-04 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Interleukine 17 (IL-17) releasing from periodontitis and peri-implantitis gingival samples | 24 hours of incubation
  Interleukine 17 (IL-17) releasing in the medium from harvested granulation tissue from periodontitis, peri-implantitis and healthy patients will be determine by ELISA test 24 hours after the beginning of the culture.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hospital Charles Foix APHP, Ivry-sur-Seine
  - Hospital Rotschild, Paris